CLINICAL TRIAL: NCT04545307
Title: Transplantation of Allogeneic Mesenchymal Stromal Cells in Patients With Immature Apex Teeth With Pulp Necrosis and Chronic Apical Periodontitis
Brief Title: Transplantation of Allogeneic MSC in Patients With Pulp Necrosis and Chronic Apical Periodontitis
Acronym: MSC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad Central de Venezuela (Other)
Collaborators: Instituto Venezolano de Investigaciones Cientificas (Other)
Responsible Party: Principal Investigator, Jose Francisco Gomez-Sosa, DDS, PhD, Instituto Venezolano de Investigaciones Cientificas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSCYPPNAP001
Record Dates: First submitted 2020-09-03; First posted 2020-09-11 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Pulp Necroses; Apical Periodontitis
Keywords: BM-MSC; Pulp regeneration
MeSH Terms: conditions — Dental Pulp Necrosis; Periapical Periodontitis

STUDY DESIGN:
Intervention Model Description: PRP clot loaded of BM-MSC in order to regenerate dental pulp tissue, placed in the root canal of an immature tooth from a patient with pulp necrosis and chronic apical periodontitis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogenic transplant of BM-MSCs (Experimental): Under sterile conditions, the patient will be locally anesthetized in the affected tooth area; the root canal of the affected tooth will be exposed and prepared to perform the MSC / MSC-Endo / PRP implant. At the same time, the culture medium supernatant is removed from each tube and the MSC / MSC-Endo "button (pellet)" is resuspended in autologous platelet-rich plasma (PRP). Subsequently to the MSC / MSC-Endo / PRP suspension, 5% CaCl2 and thrombin will be added. Immediately, and before the clot forms, 20 microliters of the MSC / MSC-Endo / PRP suspension will be placed in the root canal, covered with a collagen membrane. Subsequently, the obturation procedure with bioceramics will be carried out at the level of the pulp chamber, ionomeric glass to protect the bioceramic and later composite resin to restore the tooth.
  Interventions: Biological: Allogenic transplant of BM-MSC in a root canal from patients with immature apexes and pulpar necrosis and apical periodontitis

INTERVENTIONS:
Biological: Allogenic transplant of BM-MSC in a root canal from patients with immature apexes and pulpar necrosis and apical periodontitis — The implant of BM-MSC/MSC-Endo/PRP in a clean and shaped root canal from patients with immature apexes and pulpal necroses and apical periodontitis

SUMMARY:
The purpose of the study is to evaluate the effect of Mesenchymal Stromal Cell (MSC) implantation on pulp and periapical regeneration of immature teeth with pulp necrosis and chronic apical periodontitis.

BACKGROUND:

* Post-traumatic pulp necrosis prevents root development in children and adolescents.
* The multipotent ability of MSC to differentiate into bone-forming cells (osteoblasts) and dentin-forming cells (Odontoblast) has allowed the development of protocols to induce dental pulp regeneration in preclinical models and patients with immature teeth with pulpal necrosis.

IMPACT:

* Worldwide, post-traumatic pulp necrosis in children and adolescents constitutes a health problem in the endodontic area.
* Treatment with MSC would provide an effective therapeutic alternative to patients with pulp necrosis and incomplete root formation.
* The possible pulp and periapical regeneration of immature teeth induced by MSC would have a huge impact on the treatment of these patients.

Eligibility for EMC implant study Age: 6 to 16 years Sex: Male or Female Healthy volunteers accepted: NO.

TREATMENT GROUPS:

In the present study, the implantation of MSC will be performed in patients with immature teeth with pulpal necrosis with apical periodontitis, who will receive the appropriate endodontic treatment (according to the guidelines of the American Association of Endodontics) and implantation of allogeneic BM-MSC . This group will be compared with the history made in the Postgraduate Endodontics of the Universidad Central de Venezuela (UCV) and with international case series made by revascularization.

Clinical follow-up of each patient:

1. Clinical controls (facial evaluation, gingival evaluation, apical palpation, horizontal and vertical percussion, cold and heat sensitivity tests) will be carried out on days 0, 7, 30, 90, 180 and 364. Additionally, a clinical evaluation will be carried out at the two years post-implantation of MSC.
2. Radiological controls will be carried out on days 0, 7, 30, 90, 180 and 364. Additionally, they will be carried out two years post-implantation of MSC.
3. A tomographic evaluation will be performed when was evident periapical repair in a periapical radiograph. To measure root formation, root canal narrowing and verification the periapical repair in 3D.

DETAILED DESCRIPTION:
The endodontic procedure in the patients included in this study will focus on cases of pulp necrosis with apical periodontitis without evidence of infectious processes.

MATERIALS AND METHODS. Reagents Murine monoclonal antibodies, directed against human differentiation antigens (CD34, CD45, CD14, CD90, CD73, CD29, CD49b, CD166), conjugated to fluorescein isothiocyanate (CFI) or phycoerythrin (PE) were purchased from BD Biosciences (USA).

Isolation and culture of mesenchymal stromal cells (MSC) obtained from human bone marrow. In the present study, isolated EMFs from bone marrow (BM) from patients with a diagnosis of post-traumatic nonunion (failure of a bone union at fracture sites) will be used. These cells were transplanted into the pseudoarthrosis site to induce bone regeneration in these patients. The protocol for bone regeneration through EMF transplantation was carried out at the University Hospital of Caracas, Hospital Universitario de Los Andes, Hospital Pérez de León II and has the approval of the Bioethics Committees of each institution and each patient through informed consent. In this protocol, the BM of each patient was isolated by a puncture in the iliac crest. This procedure was performed in the operating room, under anesthesia and by a medical specialist. The MO aspirate was placed in alpha-MEM medium (Invitrogen, USA) with heparin (Sanofi Aventis). The mononuclear cells were separated by centrifugation on a Ficoll-Hypaque gradient (GE Healthcare, Sweden) and cultured in alpha-MEM-Chang medium (Irvine Scientific, USA) enriched with 20% autologous serum. These cells were kept in culture in a controlled environment at 37ºC and 5% CO2. After 72 hours, non-adherent cells were eliminated, and a basal culture medium (alpha-MEM-Chang / 20% autologous serum) was added. Their adherence to the plastic isolated the MSCs. Culture medium exchanges were made until reaching a confluence close to 70-80%. The MSCs were expanded by pealing the cultures, following the process described above. Microbiological examinations were performed after obtaining the BM and before performing the MSC implantation. After using MSC, a batch of these cells were cryopreserved at -70 -C.

Phenotypic characterization of MSC. Phenotypic characterization studies of MSC were carried out by flow cytometry. For which the MO adherent cells were detached from the culture flask by using trypsin-like enzymes. Subsequently, the cells were incubated with antibodies specific for MSC markers (CD90, CD73, CD105, CD29, CD166 and CD49b) and hematopoietic (CD34, CD45 and CD14). Cytometric analysis of the expression markers showed that 100% of the cells used for transplantation in each patient were MSC.

MSC differentiation studies. The multipotential differentiation capacity of MSCs was examined by culturing these cells in osteogenic, chondrogenic and adipogenic differentiation media, following a methodology similar to that previously described. Briefly, the MSCs were detached and seeded in 24-well culture plates at a cell density of 5x104 per well, proceeding to add the corresponding differentiation medium. For osteogenic differentiation, MSCs were cultured in the presence of basal medium enriched with dexamethasone (100nM, Biotech), ascorbic acid (10mM, Sigma), inorganic phosphate (1.8mM, Merck) and beta-glycerol phosphate (2mM, Sigma). For chondrogenic differentiation, cells were cultured in a commercial medium for chondrocytes (Cell Application, USA) and for differentiation towards the adipogenic lineage the commercial medium NH Adipodiff Human (Miltenyi, USA) was used. In all cases, the cells were kept in culture for 21-28 days with medium changes every 4-5 days. To demonstrate the changes associated with the differentiation process, the cells were fixed using paraformaldehyde (Merck, USA) and specific stains were performed for each case. Briefly, alizarin red to detect calcium deposition (evidence of osteogenesis), Alcian blue to detect proteoglycans (evidence of chondrogenesis), and oil red (Oil Red) to see lipids (evidence of adipogenesis). In all cases, microscopic observation and photographic registration were carried out. For endothelial differentiation (CEn), EMFs were cultured in MCDB 131 medium (Invitrogen, USA) enriched with 10% autologous serum, 10µg / ml of human epidermal growth factor (hu-EGF, R&D) and hydrocortisone (1µg / ml, Sigma).

MSC implantation in patients with pulp necrosis and apical periodontitis. All MSC processing procedures will be carried out in the cleanroom of the IVIC Cell Therapy Unit following the standards of good manufacturing practice (GMP). Allogeneic BM-MSC from patients diagnosed with post-traumatic nonunion and treated with implantation of these cells will be used to induce bone regeneration. The MSC to be used in this protocol have previously been phenotypically and functionally characterized. The MSC will be thawed, grown and expanded as previously described. A part of the cells will be kept in a medium for MSCs, and another part will be cultured in endothelial differentiation medium (CEM-Endo). Once the required number of MSCs and MSCs-Endo have been reached, a suspension of these cells (75,000 cells from each of them) will be placed in sterile culture tubes containing DMEM-F12 culture medium, without phenol red, supplemented with 20% autologous serum. Each tube containing MSC / MSC-Endo will be transported in a small biological sample transport cellar, at room temperature, to the Dentistry Service of the Instituto Venezolano de Investigaciones Científicas (IVIC).

Under sterile conditions, the patient will be locally anesthetized in the affected tooth area; the root canal of the affected tooth will be exposed and prepared to perform the MSC / MSC-Endo / PRP implant. At the same time, the culture medium supernatant is removed from each tube and the CEM / CEM-Endo "button (pellet)" is resuspended in autologous platelet-rich plasma (PRP). Subsequently to the MSC / Endo / PRP suspension, 5% CaCl2 and thrombin will be added. Immediately, and before the clot forms, 20 microliters of the CEM / CEM-Endo / PRP suspension will be placed in the root canal, covered with a collagen membrane. Subsequently, the obturation procedure with bioceramics will be carried out at the level of the pulp chamber, ionomeric glass to protect the bioceramic and later composite resin to restore the tooth.

Post-implantation clinical evaluation of EMF

1. Clinical controls (facial evaluation, gingival evaluation, apical palpation, horizontal and vertical percussion, cold and heat sensitivity tests) will be carried out on days 0, 7, 30, 90, 180 and 364. Additionally, a clinical evaluation will be carried out at the two years post-implantation of EMC.
2. Radiological controls will be carried out on days 0, 7, 30, 90, 180 and 364. Additionally, they will be carried out two years post-implantation of mesenchymal stromal cells.
3. A tomographic evaluation will be performed when the periapical repair will be evident in a periapical radiograph.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pulp necrosis and apical periodontitis in teeth with immature apices.
* Informed consent by the patient's representative and consent by the patient to receive bone marrow allogeneic mesenchymal stromal cell transplantation treatment.

Exclusion Criteria:

* HIV positive
* Hepatitits B or C positive
* Autoimmune diseases: lupus, rheumatoid arthritis.
* Neoplastic diseases.
* Major metabolic disorders
* Pregnancy
* Being on steroid treatment
* Other criteria that the researchers consider inappropriate for the inclusion of the patient

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Sings and Symptoms Absence | 15 days post implant
  Through clinical inspection evaluate absence of fistula, intra or extra oral inflammation, no tender to percussion or a palpation
Root canal Narrowing | 6 to 12 months
  Through periodical radiographs measure the root canal lumen months after months to evaluate any reduction of the lumen
Elongation of the root | 6 to 12 month
  Through periodical radiographs measure the teeth length from the incisal border to the apex month after month to evaluate any increase of the root length
Sensitivity tests perception | 6 to 12 months
  With the aid of pulpometer and Endo Ice evaluate if the patient start to feel any stimulation
Repair of the bone lesion produced by the apical periodontitis | 12 to 24 months
  Through a periodical radiograph evaluate month after month the increase of radiopacity in the radiolucent area produced by the apical periodontitis. When an evident repair is confirmed a tomography study will be carry out to evaluate it in 3D

SECONDARY OUTCOMES:
Stability of bio ceramic cements used in the obturation of the access cavity | 6 to 12 months
  Through periapical radiographs evaluate the maintenance of the bio ceramic cement in contact with the implant
Evaluate blood circulation within the root canal | 6 to 24 months
  By means of pulse oximeter evaluate the increase of the activity

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Terapia Celular del Instituto de Investigaciones Científicas, San Antonio de Los Altos, Miranda, Venezuela

IPD SHARING:
Plan to Share IPD: Undecided
Possibly we can share the individual clinical, radiograph and tomographic outcome of every patient enrolled in the study, mainly focus on the difficulty that every patient present.

REFERENCES:
- [Background] Antunes LS, Salles AG, Gomes CC, Andrade TB, Delmindo MP, Antunes LA. The effectiveness of pulp revascularization in root formation of necrotic immature permanent teeth: A systematic review. Acta Odontol Scand. 2016;74(3):161-9. doi: 10.3109/00016357.2015.1069394. Epub 2015 Jul 15. PMID 26179397
- [Background] Caplan AI, Dennis JE. Mesenchymal stem cells as trophic mediators. J Cell Biochem. 2006 Aug 1;98(5):1076-84. doi: 10.1002/jcb.20886. PMID 16619257
- [Background] Diaz-Solano D, Wittig O, Mota JD, Cardier JE. Isolation and Characterization of Multipotential Mesenchymal Stromal Cells from Congenital Pseudoarthrosis of the Tibia: Case Report. Anat Rec (Hoboken). 2015 Oct;298(10):1804-14. doi: 10.1002/ar.23198. Epub 2015 Jul 30. PMID 26194170
- [Background] Eramo S, Natali A, Pinna R, Milia E. Dental pulp regeneration via cell homing. Int Endod J. 2018 Apr;51(4):405-419. doi: 10.1111/iej.12868. Epub 2017 Nov 7. PMID 29047120
- [Background] Fouad AF. Microbiological aspects of traumatic injuries. Dent Traumatol. 2019 Dec;35(6):324-332. doi: 10.1111/edt.12494. Epub 2019 Oct 14. PMID 31125490
- [Background] Guerrero F, Mendoza A, Ribas D, Aspiazu K. Apexification: A systematic review. J Conserv Dent. 2018 Sep-Oct;21(5):462-465. doi: 10.4103/JCD.JCD_96_18. PMID 30294103
- [Background] Hawryluk GW, Mothe A, Wang J, Wang S, Tator C, Fehlings MG. An in vivo characterization of trophic factor production following neural precursor cell or bone marrow stromal cell transplantation for spinal cord injury. Stem Cells Dev. 2012 Aug 10;21(12):2222-38. doi: 10.1089/scd.2011.0596. Epub 2012 Feb 7. PMID 22085254
- [Background] Huang GT. Dental pulp and dentin tissue engineering and regeneration: advancement and challenge. Front Biosci (Elite Ed). 2011 Jan 1;3(2):788-800. doi: 10.2741/e286. PMID 21196351
- [Background] Iohara K, Nakashima M, Ito M, Ishikawa M, Nakasima A, Akamine A. Dentin regeneration by dental pulp stem cell therapy with recombinant human bone morphogenetic protein 2. J Dent Res. 2004 Aug;83(8):590-5. doi: 10.1177/154405910408300802. PMID 15271965
- [Background] Moradi S, Talati A, Forghani M, Jafarian AH, Naseri M, Shojaeian S. Immunohistological Evaluation of Revascularized Immature Permanent Necrotic Teeth Treated by Platelet-Rich Plasma: An Animal Investigation. Cell J. 2016 Fall;18(3):389-96. doi: 10.22074/cellj.2016.4567. Epub 2016 Aug 24. PMID 27602321
- [Background] Murakami M, Hayashi Y, Iohara K, Osako Y, Hirose Y, Nakashima M. Trophic Effects and Regenerative Potential of Mobilized Mesenchymal Stem Cells From Bone Marrow and Adipose Tissue as Alternative Cell Sources for Pulp/Dentin Regeneration. Cell Transplant. 2015;24(9):1753-65. doi: 10.3727/096368914X683502. Epub 2014 Jul 30. PMID 25199044
- [Background] Nakashima M, Iohara K. Regeneration of dental pulp by stem cells. Adv Dent Res. 2011 Jul;23(3):313-9. doi: 10.1177/0022034511405323. PMID 21677085
- [Background] Pittenger MF, Mackay AM, Beck SC, Jaiswal RK, Douglas R, Mosca JD, Moorman MA, Simonetti DW, Craig S, Marshak DR. Multilineage potential of adult human mesenchymal stem cells. Science. 1999 Apr 2;284(5411):143-7. doi: 10.1126/science.284.5411.143. PMID 10102814
- [Background] Shammaa R, El-Kadiry AE, Abusarah J, Rafei M. Mesenchymal Stem Cells Beyond Regenerative Medicine. Front Cell Dev Biol. 2020 Feb 18;8:72. doi: 10.3389/fcell.2020.00072. eCollection 2020. PMID 32133358
- [Background] Wang X, Thibodeau B, Trope M, Lin LM, Huang GT. Histologic characterization of regenerated tissues in canal space after the revitalization/revascularization procedure of immature dog teeth with apical periodontitis. J Endod. 2010 Jan;36(1):56-63. doi: 10.1016/j.joen.2009.09.039. PMID 20003936
- [Background] Wittig O, Diaz-Solano D, Cardier J. Viability and functionality of mesenchymal stromal cells loaded on collagen microspheres and incorporated into plasma clots for orthopaedic application: Effect of storage conditions. Injury. 2018 Jun;49(6):1052-1057. doi: 10.1016/j.injury.2018.04.005. Epub 2018 Apr 5. PMID 29678307
- [Background] Wittig O, Romano E, Gonzalez C, Diaz-Solano D, Marquez ME, Tovar P, Aoun R, Cardier JE. A method of treatment for nonunion after fractures using mesenchymal stromal cells loaded on collagen microspheres and incorporated into platelet-rich plasma clots. Int Orthop. 2016 May;40(5):1033-8. doi: 10.1007/s00264-016-3130-6. Epub 2016 Mar 16. PMID 26980620
- [Background] Xuan K, Li B, Guo H, Sun W, Kou X, He X, Zhang Y, Sun J, Liu A, Liao L, Liu S, Liu W, Hu C, Shi S, Jin Y. Deciduous autologous tooth stem cells regenerate dental pulp after implantation into injured teeth. Sci Transl Med. 2018 Aug 22;10(455):eaaf3227. doi: 10.1126/scitranslmed.aaf3227. PMID 30135248